CLINICAL TRIAL: NCT02142361
Title: Clinical Performance of Habitual Wearers of Hydrogel Toric Lenses When Refitted With Avaira Toric Silicone Hydrogel Lenses
Brief Title: Clinical Performance of Habitual Hydrogel vs. Silicone Hydrogel Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EX-MKTG-48
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Results first posted 2016-04-19 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Omafilcon A/Enfilcon A (Active Comparator): Subject's habitual hydrogel toric lenses Omafilcon A will be evaluated at the first visit and then re-fitted with a pair of Enfilcon A lenses.
  Interventions: Device: enfilcon A
- Ocufilcon D/Enfilcon A (Active Comparator): Subject's habitual hydrogel toric lenses Ocufilcon D will be evaluated at the first visit and then re-fitted with a pair of Enfilcon A lenses.
  Interventions: Device: enfilcon A
- Methafilcon B/ Enfilcon A (Active Comparator): Subject's habitual hydrogel toric lenses Methafilcon B will be evaluated at the first visit and then re-fitted with a pair of Enfilcon A lenses.
  Interventions: Device: enfilcon A

INTERVENTIONS:
Device: enfilcon A — Silicone hydrogel toric lenses.
  Other Names: enfilcon A/Silicone Hydrogel Lens

SUMMARY:
Evaluate the clinical performance of existing wearers of hydrogel toric lenses when refitted with Avaira toric silicone hydrogel contact lenses over 1 week of wear.

DETAILED DESCRIPTION:
This is a 60-subject, single masked, bilateral, parallel study design comparing the fitting characteristics of enfilcon A toric lenses against the subjects habitual hydrogel toric lenses (omafilcon A, ocufilcon D or methafilcon B wearers). Subject's habitual toric lenses will be evaluated at the first visit and then re-fitted with a pair of Avaira toric lenses. After 1 week of daily wear, subjects will return for a second and final evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 40 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Is an adapted soft toric contact lens wearer
* Has a contact lens spherical prescription between +6.00 to - 8.00 (inclusive)
* Have no less than 0.75D of astigmatism and no more than 1.75 D in both eyes.
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter.
* Patient contact lens refraction should fit within the available parameters of the study lenses.
* Is willing to comply with the wear schedule (at least 5 days per week, > 8 hours/day assuming there are no contraindications for doing so).
* Is willing to comply with the visit schedule

Exclusion Criteria:

* Has a contact lens prescription outside the range of the available parameters of the study lenses.
* Has a spectacle cylinder less than -0.75D or more than -1.75D of cylinder in either eye.
* Has a history of not achieving comfortable contact lens wear (5 days per week; > 8 hours/day)
* Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye.
* Presence of clinically significant (grade 2-4) anterior segment abnormalities
* Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear such as:

  * Pathological dry eye or associated findings
  * Pterygium, pinguecula, or corneal scars within the visual axis
  * Neovascularization > 0.75 mm in from of the limbus
  * Giant papillary conjunctivitis (GCP) worse than grade 1
  * Anterior uveitis or iritis (past or present)
  * Seborrheic eczema, Seborrheic conjunctivitis
  * History of corneal ulcers or fungal infections
  * Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea.
* Has Presbyopia or has dependence on spectacles for near work over the contact lenses.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Montés-Mico, OD MPhil PhD, Principal Investigator — Optometry Research Group (GIO) Optics Department, University of Valencia
Locations (1):
- Optometry Research Group (GIO) Optics Department, University of Valencia, Valencia, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- Omafilcon A/Enfilcon A: Subject's habitual hydrogel toric lenses (omafilcon A) will be evaluated at the first visit and then re-fitted with a pair of silicon hydrogel toric lenses (enfilcon A).
- Ocufilcon D/Enfilcon A: Subject's habitual hydrogel toric lenses (ocufilcon D) will be evaluated at the first visit and then re-fitted with a pair of silicon hydrogel toric lenses (enfilcon A).
- Methafilcon B/Enfilcon A: Subject's habitual hydrogel toric lenses (methafilcon B) will be evaluated at the first visit and then re-fitted with a pair of silicon hydrogel toric lenses (enfilcon A).
Period: Overall Study
Arm/Group | Omafilcon A/Enfilcon A | Ocufilcon D/Enfilcon A | Methafilcon B/Enfilcon A
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The subject sample consisted of 60 habitual hydrogelcontact lens wearers (omafilcon A, ocufilcon D or methafilcon B), refitted with silicone hydrogel lens (enfilcon A)
Groups:
- Overall Study Group: All participants were habitual wearers of hydrogel toric lenses (omafilcon A, ocufilcon D or methafilcon B), and refitted with silicone hydrogel toric lens (enfilcon A)
Arm/Group | Overall Study Group
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Participant's Subjective Rating for Lens Initial Comfort
Description: Surveyed for habitual pair at baseline. Dispensed pair after insertion/settling at 1 week. Rated on a visual analog scale (VAS). (0-10, 0=poor, 10= can't feel)
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Omafilcon A: Subject's habitual hydrogel toric lenses (omafilcon A) will be evaluated at the first visit and then re-fitted with a pair of silicon hydrogel toric lenses (enfilcon A).
- Ocufilcon D: Subject's habitual hydrogel toric lenses (ocufilcon D) will be evaluated at the first visit and then re-fitted with a pair of silicon hydrogel toric lenses (enfilcon A).
- Methafilcon B: Subject's habitual hydrogel toric lenses (methafilcon B) will be evaluated at the first visit and then re-fitted with a pair of silicon hydrogel toric lenses (enfilcon A).
Arm/Group | Omafilcon A | Ocufilcon D | Methafilcon B
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Habitual lens-Baseline | 6.9 (1.4) | 7.4 (1.3) | 8.0 (1.1)
  Study lens-1 Week | 8.9 (1.3) | 7.8 (1.8) | 8.1 (1.7)

2. Primary Outcome: Participant's Subjective Rating for Lens Comfort Prior to Removal
Description: Surveyed prior to removal of each lens pair. Habitual pair at baseline. Dispensed pair at 1 week. Rated on a visual analog scale (VAS). (0-10, 0=poor, 10= can't feel)
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Ocufilcon D | Methafilcon B
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Habitual lens -Baseline | 7.4 (1.2) | 7.4 (1.7) | 6.7 (2.0)
  Study Lens -1 week | 8.2 (1.4) | 8.0 (1.4) | 7.3 (2.3)

3. Primary Outcome: Participant's Subjective Rating for Overall Lens Comfort
Description: Surveyed for each lens pair. Habitual pair at baseline. Dispensed pair at 1 week. Rated on a visual analog scale (VAS). (0-10, 0=poor, 10= can't feel)
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Ocufilcon D | Methafilcon B
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Habitual lens- Baseline | 8.2 (1.1) | 8.4 (1.0) | 8.2 (1.2)
  Study lens-1 week | 8.8 (1.1) | 8.4 (1.2) | 8.4 (1.4)

4. Primary Outcome: Participant's Subjective Rating for Dryness During the Day
Description: Surveyed for each lens pair. Habitual pair at baseline. Dispensed pair at 1 week. Rated on a visual analog scale (VAS). (0-10, 0=very dry, 10= no dryness)
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Ocufilcon D | Methafilcon B
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Habitual lens-Baseline | 7.7 (1.5) | 8.0 (0.9) | 7.4 (1.7)
  Study lens-1 week | 8.6 (1.5) | 8.1 (1.6) | 8.2 (1.6)

5. Primary Outcome: Participant's Subjective Rating for Dryness Prior to Removal
Description: Surveyed prior to removal of each lens pair. Habitual pair at baseline . Dispensed pair at 1 week. Rated on a visual analog scale (VAS). (0-10, 0=very dry, 10= no dryness)
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Ocufilcon D | Methafilcon B
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Habitual lens-Baseline | 7.4 (1.4) | 7.0 (1.3) | 6.3 (2.2)
  Study lens-1 week | 7.7 (1.7) | 7.5 (1.9) | 7.5 (2.1)

6. Primary Outcome: Participant's Subjective Rating for Overall Dryness
Description: Surveyed for each lens pair. Habitual pair at baseline. Dispensed pair at 1 week . Rated on a visual analog scale (VAS). (0-10, 0=very dry, 10= no dryness)
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Ocufilcon D | Methafilcon B
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Habitual lens-Baseline | 7.8 (1.3) | 7.6 (1.0) | 7.2 (1.9)
  Study lens-1 week | 8.8 (1.2) | 8.3 (1.4) | 8.2 (1.7)

7. Primary Outcome: Participant's Subjective Rating for Lens Handling - Insertion
Description: Surveyed for habitual pair at baseline. Dispensed pair after insertion/settling at 1 week. Rated on a visual analog scale (VAS). (0-10, 0=poor, 10= very easy)
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Ocufilcon D | Methafilcon B
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Habitual lens-Baseline | 8.4 (1.2) | 8.8 (1.4) | 9.1 (0.8)
  Study lens-1 week | 9.3 (0.7) | 8.8 (1.0) | 9.5 (0.9)

8. Primary Outcome: Participant's Subjective Rating for Overall Lens Fit Stability
Description: Surveyed for each lens pair. Habitual pair at baseline. Dispensed pair at 1 week. Rated on a visual analog scale (VAS). (0-10, 0=very unstable / excessive movement, 10= very stable / good movement)
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Ocufilcon D | Methafilcon B
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Habitual lens-Baseline | 8.1 (1.3) | 7.8 (1.5) | 7.9 (1.7)
  Study Lens- 1 week | 8.1 (1.8) | 8.0 (1.5) | 9.0 (0.8)

9. Primary Outcome: Participant's Subjective Rating for Overall Vision Satisfaction
Description: Surveyed for each lens pair. Habitual pair at baseline. Dispensed pair at 1 week. Rated on a visual analog scale (VAS). (0-10, 0=completely dissatisfied, 10= very satisfied)
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Ocufilcon D | Methafilcon B
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Habitual lens- Baseline | 8.3 (1.1) | 8.1 (1.6) | 8.6 (1.4)
  Study lens-1 week | 8.6 (1.1) | 8.7 (1.0) | 9.3 (0.7)

10. Primary Outcome: Participant's Subjective Rating for Vision Quality at Insertion
Description: Surveyed for habitual pair at baseline. Dispensed pair after insertion/settling at 1 week .Rated on a visual analog scale (VAS). (0-100, 0=extremely poor vision totally blurred, 100= excellent vision totally sharp)
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Ocufilcon D | Methafilcon B
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Habitual lens-Baseline | 77 (10.3) | 75.5 (11.9) | 79.5 (10.0)
  Study lens-1 week | 87.5 (12.1) | 82.5 (12.5) | 86.5 (9.3)

11. Primary Outcome: Participant's Subjective Rating for Vision Quality During the Day
Description: Surveyed for each lens pair. Habitual pair at baseline. Dispensed pair at 1 week . Rated on a visual analog scale (VAS). (0-100, 0=extremely poor vision totally blurred, 100= excellent vision totally sharp)
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Ocufilcon D | Methafilcon B
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Habitual lens-Baseline | 83 (11.3) | 86 (11.0) | 84.5 (11.9)
  Study lens-1 week | 87.5 (11.2) | 85 (8.9) | 91.5 (7.5)

12. Primary Outcome: Participant's Subjective Rating for Vision Quality End of the Day
Description: Surveyed for each lens pair. Habitual pair at baseline. Dispensed pair at 1 week end of the day. Rated on a visual analog scale (VAS). (0-100, 0=extremely poor vision totally blurred, 100= excellent vision totally sharp)
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Ocufilcon D | Methafilcon B
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Habitual lens-Baseline | 79 (10.2) | 82.5 (14.1) | 76 (14.1)
  Study lens-1 week | 79.8 (17.2) | 80.5 (13.9) | 87.5 (9.7)

13. Primary Outcome: Participant's Subjective Rating for Night Vision Quality
Description: Surveyed for each lens pair. Habitual pair at baseline. Study pair dispensed pair at 1 week. Rated on a visual analog scale (VAS). (0-100, 0=extremely poor vision totally blurred, 100= excellent vision totally sharp)
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Ocufilcon D | Methafilcon B
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Habitual lens-Baseline | 77.3 (7.2) | 83.3 (10.5) | 81.8 (10.0)
  Study lens-1 week | 83.5 (8.6) | 84.5 (7.8) | 87.3 (8.7)

14. Primary Outcome: Participant's Subjective Rating for Vision Stability at Insertion
Description: Surveyed for habitual pair at baseline. Dispensed pair after insertion/settling at 1 week. Rated on a visual analog scale (VAS). (0-100, 0=Totally unstable Fluctuating/changing, 100= perfectly stable Not fluctuating/changing)
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Ocufilcon D | Methafilcon B
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Habitual lenses-Baseline | 74 (10.5) | 70 (12.6) | 71.5 (15.3)
  Study lens-1 week | 86.5 (11.4) | 81 (14.1) | 85.5 (10.5)

15. Primary Outcome: Participant's Subjective Rating for Vision Stability During the Day
Description: Surveyed for each lens pair. Habitual pair at baseline. Dispensed pair at 1 week. Rated on a visual analog scale (VAS). (0-100, 0=Totally unstable Fluctuating/changing, 100= perfectly stable Not fluctuating/changing)
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Ocufilcon D | Methafilcon B
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Habitual lens-Baseline | 83 (8.6) | 81.5 (10.9) | 77.5 (16.2)
  Study lens-1 week | 82.5 (11.6) | 82.5 (12.1) | 90 (7.9)

16. Primary Outcome: Participant's Subjective Rating for Vision Stability at End of Day
Description: as for outcome 15
Time Frame: Baseline and 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omafilcon A | Ocufilcon D | Methafilcon B
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Habitual lens-Baseline | 81 (9.1) | 79.5 (13.9) | 75.5 (16.4)
  Study lens-1 week | 77.5 (16.8) | 82 (13.2) | 88.5 (7.5)

17. Primary Outcome: Participant's Subjective Rating for Lens Pair Preference
Description: Participants subjective preference in relation to comfort, dryness, handling, vision, lens fit and overall of the patient after wearing the study and their habitual lenses.
Time Frame: 1 week
Population: All 60 paticipants were analyzed for the habitual lenses. The results have been combined into a single arm "Habitual Lens" arm to create a single pair wise comparison to the, "Study Lens" arm. "Vision" category data for one participant was not collected.
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: eyes
Groups:
- Habitual Lenses: Subjects habitual hydrogel toric lens pairs surveyed at 1 week.
- Study Lens: Subjects dispensed with study lens pair (Enfilcon A) pair and surveyed 1 week.
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (eyes) | 120 | 120
Percentage of eyes
  Overall | 10 | 90
  Comfort | 13 | 87
  Dryness | 25 | 75
  Handling | 17 | 83
  Vision | 13 | 85
  Lens Fit | 10 | 90

18. Primary Outcome: Participant's Subjective Rating for Overall Satisfaction - Dryness
Description: Surveyed for each lens pair. Habitual pair at baseline. Dispensed pair at 1 week . Likert scale. (4 choices - completely satisfied, somewhat satisfied, somewhat dissatisfied, completely dissatisfied)
Time Frame: Baseline and 1 week
Population: All 60 participants were analyzed for the habitual lenses. The results have been combined into a single arm "Habitual Lens" arm to create a single pair wise comparison to the, "Study Lens" arm.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Groups:
- Habitual Lenses: Subjects habitual hydrogel toric lens pairs surveyed at baseline.
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  completely satisfied | 27 | 40
  somewhat satisfied | 55 | 42
  somewhat dissatisfied | 18 | 13
  completely dissatisfied | 0 | 5

19. Primary Outcome: Participant's Subjective Rating for Overall Satisfaction - Handling
Description: as for outcome 18
Time Frame: Baseline and 1 week
Population: All 60 participants were analyzed for the habitual lenses. The results have been combined into a single arm "Habitual Lens" arm to create a single pair wise comparison to the, "Study Lens" arm.
  Sum of percentage for the Study Lens Arm=101 as, Category title- " Somewhat dissatisfied- 1.7 was rounded to 2.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  completely satisfied | 73 | 87
  somewhat satisfied | 23 | 12
  somewhat dissatisfied | 3 | 2
  completely dissatisfied | 0 | 0

20. Primary Outcome: Participant's Subjective Rating for Overall Satisfaction - Vision
Description: as for outcome 18
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  completely satisfied | 48 | 62
  somewhat satisfied | 43 | 37
  somewhat dissatisfied | 8 | 0
  completely dissatisfied | 0 | 0

21. Primary Outcome: Participant's Subjective Rating for Overall Satisfaction - Lens Fit
Description: Surveyed for each lens pair. Habitual pair at baseline. Dispensed pair at 1 week. Likert scale. (4 choices - completely satisfied, somewhat satisfied, somewhat dissatisfied, completely dissatisfied)
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  completely satisfied | 40 | 65
  somewhat satisfied | 42 | 23
  somewhat dissatisfied | 18 | 12
  completely dissatisfied | 0 | 0

22. Primary Outcome: Participant's Subjective Rating for Overall Satisfaction - Overall
Description: as for outcome 21
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  completely satisfied | 30 | 58
  somewhat satisfied | 67 | 42
  somewhat dissatisfied | 3 | 0
  completely dissatisfied | 0 | 0

23. Primary Outcome: Clinician's Objective Assessment Monocular High Contrast Distance Visual
Description: Assessed for each lens pair. Habitual pair at baseline. Dispensed pair at 1 week. LogMAR - Positive values denote poorer vision, negative values denote better vision than baseline 20/20 value.
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
LogMAR
  VA Oculus Dexter (OD) | -0.037 (0.049) | -0.037 (0.049)
  VA Oculus Sinister (OS) | -0.037 (0.049) | -0.037 (0.049)

24. Primary Outcome: Clinician's Objective Assessment Binocular High Contrast Distance Visual Acuity
Description: as for outcome 23
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
LogMAR | -0.037 (0.0049) | -0.037 (0.0049)

25. Primary Outcome: Clinician's Assessment Overall Lens Stability-Right Eye
Description: Surveyed for habitual pair at baseline. Dispensed pair after insertion/settling at 1 week. Overall performance of the lens in terms of axis stability on primary gaze, during lateral gaze, rotational recovery, and mislocation of the lens on blinking. Likert scale. (0-4, 0=very poor,1=poor, 2=moderate, 3=good, 4= excellent)
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 60 | 60
percentage of eyes
  Very Poor | 0 | 0
  Poor | 0 | 0
  Moderate | 0 | 0
  Good | 62 | 8
  Excellent | 38 | 92

26. Primary Outcome: Clinician's Assessment Overall Lens Stability-Left Eye
Description: as for outcome 25
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 60 | 60
percentage of eyes
  Very Poor | 0 | 0
  Poor | 0 | 0
  Moderate | 0 | 0
  Good | 55 | 5
  Excellent | 45 | 95

27. Primary Outcome: Clinician's Assessment Overall Fit Acceptance- Right Eye
Description: Surveyed for habitual pair at baseline. Dispensed pair after insertion/settling at 1 week. Overall fit acceptance based on lens fit alone (not comfort or vision). Likert scale. (0-4, 0=Very poor 1=Poor 2=Moderate, 3=Good, 4= Excellent)
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 60 | 60
percentage of eyes
  Very Poor | 0 | 0
  Poor | 0 | 0
  Moderate | 0 | 0
  Good | 48 | 3
  Excellent | 52 | 97

28. Primary Outcome: Clinician's Assessment Overall Fit Acceptance- Left Eye
Description: as for outcome 27
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 60 | 60
percentage of eyes
  Very Poor | 0 | 0
  Poor | 0 | 0
  Moderate | 0 | 0
  Good | 48 | 3
  Excellent | 52 | 97

29. Primary Outcome: Clinician's Assessment Lens Centration-Right Eye
Description: Surveyed for habitual pair at baseline. Dispensed pair after insertion/settling at 1 week . Lens centration recorded by degree and direction in the primary position. (0-2, 0=centered/optimal, 1=decentered slightly, 2=substantially decentered (>0.5mm))
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 60 | 60
percentage of eyes
  Centered | 100 | 100
  Slightly decentered | 0 | 0
  Substantially decentered | 0 | 0

30. Primary Outcome: Clinician's Assessment Lens Centration- Left Eye
Description: Surveyed for habitual pair at baseline. Dispensed pair after insertion/settling at 1 week. Lens centration recorded by degree and direction in the primary positions. (0-2, 0=centered/optimal, 1=decentered slightlty, 2=substantially decentered (>0.5mm)
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 60 | 60
percentage of eyes
  Centered | 100 | 100
  Slightly decentered | 0 | 0
  Substantially decentered | 0 | 0

31. Primary Outcome: Clinician's Assessment Corneal Coverage-Right Eye
Description: Surveyed for habitual pair at baseline. Dispensed pair after insertion/settling at 1 week. Assessed in primary gaze. (Y=yes, full corneal coverage at all times, N=no, incomplete corneal coverage)
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 60 | 60
percentage of eyes
  Full corneal coverage | 100 | 100
  Incomplete corneal coverage | 0 | 0

32. Primary Outcome: Clinicians Assessment Corneal Coverage-Left Eye
Description: Surveyed for habitual pair at baseline. Dispensed pair after insertion/settling at 1 week. Assessed in primary gaze. (Y=yes, full corneal coverage at all times, N=no incomplete corneal coverage)
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 60 | 60
percentage of eyes
  Full corneal coverage | 100 | 100
  Incomplete corneal coverage | 0 | 0

33. Primary Outcome: Clinician's Assessment Post-Blink Movement- Right Eye
Description: Surveyed for habitual pair at baseline. Dispensed pair after insertion/settling at 1 week. Assessed immediately after the blink. (0-4, 0=insufficient, unacceptable movement, 1=minimal, but acceptable movement, 2=optimal movement, 3=moderate, but acceptable movement, 4=excessive, unacceptable movement
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 60 | 60
percentage of eyes
  Insufficient/Unacceptable movement | 0 | 0
  Minimal, but acceptable movement | 0 | 0
  Optimal movement, | 100 | 100
  Moderate, but acceptable movement | 0 | 0
  Excessive, inacceptable movement | 0 | 0

34. Primary Outcome: Clinician's Assessment Post-Blink Movement-Left Eye
Description: as for outcome 33
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 60 | 60
percentage of eyes
  Insufficient/Unacceptable movement | 0 | 0
  Minimal, but acceptable movement | 0 | 0
  Optimal movement | 100 | 100
  Moderate, but acceptable movement | 0 | 0
  Excessive,unacceptable movement | 0 | 0

35. Primary Outcome: Clinician's Assessment Lens Orientation in Primary Position of Gaze- Right Eye
Description: Assessed for habitual pair at baseline. Dispensed pair after insertion/settling at 1 week . Slit lamp, with 10x magnification. Nasal mislocation is recorded as (+) and temporal as (-). Mislocation of the axis mark on the lens relative to the 6 o'clock position, zero rotation, measured in degrees.
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 60 | 60
percentage of eyes
  Temporal | 12 | 0
  0 rotation | 18 | 100
  Nasal | 70 | 0

36. Primary Outcome: Clinician's Assessment Lens Orientation in Primary Position of Gaze-Left Eye
Description: as for outcome 35
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 60 | 60
percentage of eyes
  Temporal | 12 | 0
  0 rotation | 73 | 100
  Nasal | 15 | 0

37. Primary Outcome: Clinician's Assessment Rotational Recovery in Degrees After 60 Seconds-Right Eye
Description: Assessed for habitual pair at baseline. Dispensed pair after insertion/settling at 1 week . Slit lamp, with 10x magnification. Lens ability to return to its original position measured 60 seconds after manually rotating the lens 45 degrees temporally.
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 60 | 60
degrees | 0 (0) | 0 (0)

38. Primary Outcome: Clinician's Assessment Rotational Recovery in Degrees After 60 Seconds-Left Eye
Description: as for outcome 37
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 60 | 60
degrees | 0 (0) | 0 (0)

39. Primary Outcome: Participant's Subjective Rating for Overall Satisfaction - Comfort
Description: as for outcome 21
Time Frame: Baseline and 1 week
Population: as for outcome 18
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Habitual Lenses | Study Lens
Number analyzed (Participants) | 60 | 60
Number analyzed (Eyes) | 120 | 120
percentage of eyes
  Completely satisfied | 30 | 55
  somewhat satisfied | 58 | 40
  somewhat dissatisfied | 12 | 5
  completely dissatisfied | 0 | 0

ADVERSE EVENTS:
Time Frame: From Dispense up to one week for each study lenses
Groups:
- Omafilcon A; Ocufilcon D; Methafilcon B: Subject's habitual hydrogel toric lenses will be evaluated at the first visit and then re-fitted with a pair of silicon hydrogel toric lenses. After 1 week of daily wear, subjects will return for a second and final evaluation.
  enfilcon A: Subject's habitual hydrogel toric lenses will be evaluated at the first visit and then re-fitted with a pair of silicon hydrogel toric lenses. After 1 week of daily wear, subjects will return for a second and final evaluation.
Arm/Group | Omafilcon A | Ocufilcon D | Methafilcon B
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study.

There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor.